CLINICAL TRIAL: NCT03061136
Title: Clonazepam Effects on Brain Oscillations and Cognition in Schizophrenia
Acronym: KGB
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Delays in equipment procurement prevented the start of the study in time
Sponsor: Palo Alto Veterans Institute for Research (Other)
Collaborators: Stanford University (Other); University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Jong Yoon, Principal Investigator, Palo Alto Veterans Institute for Research
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: YOJ0004ARC
Record Dates: First submitted 2017-02-15; First posted 2017-02-23 (Actual); Last update posted 2018-04-05 (Actual); Status verified 2018-04

CONDITIONS: Schizophrenia; Schizoaffective Disorder; Schizophreniform Disorder
Keywords: Cognition; Gamma oscillations; EEG; Executive function; Benzodiazepine; GABA
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Clonazepam

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Placebo (Placebo Comparator): Placebo administered orally
  Interventions: Drug: Placebo
- Clonazepam 0.1mg (Experimental): 0.1mg clonazepam administered orally
  Interventions: Drug: Clonazepam
- Clonazepam 0.2mg (Experimental): 0.2mg clonazepam administered orally
  Interventions: Drug: Clonazepam
- Clonazepam 0.3mg (Experimental): 0.3mg clonazepam administered orally
  Interventions: Drug: Clonazepam

INTERVENTIONS:
Drug: Clonazepam
  Other Names: Klonopin
  Arms: Clonazepam 0.1mg; Clonazepam 0.2mg; Clonazepam 0.3mg
Drug: Placebo
  Arms: Placebo

SUMMARY:
Cognitive deficits are some of the most prominent and disabling symptoms of schizophrenia. Evidence suggests that schizophrenia involves alterations to the functioning of a neural system under the control of a brain chemical called GABA. The present project will compare the effects of low-dose clonazepam (at a sub-sedating dose) to placebo, for effects on GABA- modulated brain activity measured by EEG, and associated cognitive processes in people who have schizophrenia.

DETAILED DESCRIPTION:
Schizophrenia is a common, disabling mental illness with a considerable public health impact. Cognitive dysfunction (e.g in attention, memory, etc.) is an enduring feature of the illness, a strong predictor of functional outcome, and presently has no established treatment. Therefore, advances in treatment of cognition in schizophrenia are likely to alleviate a significant health burden. Deficits in executive control functions, such as those measurable on task-switching paradigms, are among the most important cognitive deficits in schizophrenia, and arise from disturbances in distributed neural networks operated by the prefrontal cortex. An important phenomenon that underpins cortical information processing are oscillations in brain activity that can be measured both with intracranial electrical recordings and at the scalp with EEG. These networks and their cortical oscillatory signatures are also strongly modulated by cortical interneurons that use gamma-amino butyric acid (GABA) as a neurotransmitter. Post-mortem evidence suggests that GABAergic neurons are altered in schizophrenia. Furthermore, studies in animals, using optogenetic manipulations that are restricted to a subset of cortical GABA neurons, also suggest that GABA neurons can be selectively modulated to improve PFC-dependent cognition in animal models of schizophrenia. This includes experiments that involve administration of sub-sedating doses of clonazepam, a representative FDA-approved medication from the benzodiazepine class.

Therefore, this neurochemical system represents a novel set of candidate treatment targets that are both implicated in the pathophysiology of schizophrenia and the potential remediation of associated cognitive dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* Subjects will be included if they are adults (18-55 years old) who currently meet criteria for schizophrenia, schizophreniform disorder or schizoaffective disorder from the DSM-IV (295.X).
* Healthy control subjects: 18-55 years of age.

Exclusion Criteria:

* All subjects will be excluded if they have a history of any substance-related disorder (by DSM-IV, other than cannabis abuse) in the prior 6 months, or repeated positive urine drug screens for other illicit substances. They will also be excluded if they are clinically-unstable, have significant baseline or emergent suicide risk (by Columbia Suicide Severity Risk Scale), estimated IQ < 70, or EEG contraindications. Subjects must also have no major medical or neurological illness, or significant head trauma.
* Active pregnancy or lactation will also be considered contraindications for treatment with clonazepam, and as criteria for exclusion.

Excluded medications:

* Prospective subjects will be excluded if they are currently in treatment with benzodiazepines, anticonvulsants, and medications such as zolpidem and baclofen, each of which directly affect GABA neurons or may be associated with changes in GABA system function.
* Known allergy/sensitivity or any hypersensitivity to components of study drug(s) or their formulation, or sensitivity/hypersensitivity to clonazepam will be criteria for exclusion.
* Healthy controls must be free of a diagnosis of a chronic or recurrent Axis I (or certain Axis II) psychiatric disorder and will be excluded if they have a first degree relative with a psychotic disorder.
* Education, parental education, ethnicity, handedness, and native language will be used as exclusionary factors as necessary to maintain balanced groups. This information is collected during the telephone screen to ensure group balance.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2016-10; Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
EEG Gamma-oscillatory power | 1 day
  Gamma-oscillation power is derived from EEG spectrogram, reflecting underlying brain electrical activity

SECONDARY OUTCOMES:
EEG derived Auditory steady state power | 1 day
  Auditory steady state power is derived from EEG spectrogram, reflecting underlying brain electrical activity responding to auditory stimulation
Brief Psychiatric Rating Scale (BPRS) | 1 day
  Quantification of level of psychopathology, rater-administered survey
Scale for the Assessment of Negative Symptoms (SANS) | 1 day
  Quantification of level of negative symptoms, rater-administered survey
Scale for the Assessment of Positive Symptoms (SAPS) | 1 day
  Quantification of level of positive symptoms, rater-administered survey
Working memory task accuracy | 1 day
  Subject's behavioral performance on a working memory task

CONTACTS AND LOCATIONS:
Locations (1):
- VA Palo Alto Health Care System, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bowie CR, Harvey PD. Cognition in schizophrenia: impairments, determinants, and functional importance. Psychiatr Clin North Am. 2005 Sep;28(3):613-33, 626. doi: 10.1016/j.psc.2005.05.004. PMID 16122570
- [Background] Minzenberg MJ, Carter CS. Developing treatments for impaired cognition in schizophrenia. Trends Cogn Sci. 2012 Jan;16(1):35-42. doi: 10.1016/j.tics.2011.11.017. Epub 2011 Dec 16. PMID 22178120
- [Background] Lesh TA, Niendam TA, Minzenberg MJ, Carter CS. Cognitive control deficits in schizophrenia: mechanisms and meaning. Neuropsychopharmacology. 2011 Jan;36(1):316-38. doi: 10.1038/npp.2010.156. Epub 2010 Sep 15. PMID 20844478
- [Background] Minzenberg MJ, Laird AR, Thelen S, Carter CS, Glahn DC. Meta-analysis of 41 functional neuroimaging studies of executive function in schizophrenia. Arch Gen Psychiatry. 2009 Aug;66(8):811-22. doi: 10.1001/archgenpsychiatry.2009.91. PMID 19652121
- [Background] Cho KK, Hoch R, Lee AT, Patel T, Rubenstein JL, Sohal VS. Gamma rhythms link prefrontal interneuron dysfunction with cognitive inflexibility in Dlx5/6(+/-) mice. Neuron. 2015 Mar 18;85(6):1332-43. doi: 10.1016/j.neuron.2015.02.019. Epub 2015 Mar 5. PMID 25754826